CLINICAL TRIAL: NCT03665493
Title: Dopamine Effect on Inhibitory Control
Acronym: DEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giovanni Mirabella (Other)
Responsible Party: Sponsor-Investigator, Giovanni Mirabella, Principal Investigator, Neuromed IRCCS
Organization: Neuromed IRCCS (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: GMirab_01
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Levodopa medication; stop signal task; inhibitory control; Parkinson's Disease; stop signal reaction time; proactive inhibition
MeSH Terms: conditions — Parkinson Disease; Proactive Inhibition

STUDY DESIGN:
Intervention Model Description: Both groups of patients will perform the stop-signal task and the go-only task under two conditions: a) ON Levodopa medication state calculated after the first-morning dose which normally allowed the patient to attain the best control of symptoms (4) b) OFF Levodopa medication state. i.e patients did not take medications overnight prior to the study (19). Experimental conditions will be counterbalanced across patients and administered in two different experimental sessions occurring on different days.
  Healthy controls will perform the stop signal task and the go-only task in the same day. The order of administration will be counterbalanced.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PD patients H&Y=1.5-2 Medications ON (Experimental): Idiopathic Parkinson's patient's with Hoehn and Yahr score of 1.5- 2 i.e. in an early stage of the disease, under stable treatment with the administration of L-dopa and dopamine agonists. Patients will not present severe sensory deficits or any other neurological disease besides PD, as will be assessed by a standard neurological examination, and they will be all right-handed as will be assessed by the Edinburgh handedness inventory. Age range: 40-70
  Interventions: Drug: PD patients H&Y=1.5-2 Medications ON
- PD patients H&Y=3 Medications ON (Experimental): Parkinson's patient's with Hoehn and Yahr score of 3, i.e. in moderate-to-advanced stages of the disease under stable treatment with the administration of L-dopa and dopamine agonists. Patients will not present severe sensory deficits or any other neurological disease besides PD, as will be assessed by a standard neurological examination, and they will be all right-handed as will be assessed by the Edinburgh handedness inventory. Age range: 40-70
  Interventions: Drug: PD patients H&Y=3 Medications ON
- PD patients H&Y=1.5-2 Medications OFF (Experimental): Same as above described
  Interventions: Drug: PD patients H&Y=1.5-2 Medications OFF
- PD patients H&Y=3 Medications OFF (Experimental): Same as above described
  Interventions: Drug: PD patients H&Y=3 Medications OFF
- Healthy age-matched controls (Experimental): Healthy controls. Right-handed healthy subjects (it will be assessed by the Edinburgh handedness inventory) with normal or corrected-to-normal vision, without a history of neurological diseases. Age range: 40-70.
  Interventions: Behavioral: Healthy age-matched controls

INTERVENTIONS:
Drug: PD patients H&Y=1.5-2 Medications ON — Parkinson's patients will be allowed to the first-morning dose of levodopa medicament (levodopa, dopamine agonists, anticholinergic drugs, or a combination of levodopa and an anticholinergic drug) which normally allowed the patient to attain the best control of symptoms one hour before being tested (19). Patients will perform both the stop-signal task and the go-only task. Experimental conditions will be counterbalanced across patients.
  Arms: PD patients H&Y=1.5-2 Medications ON
Drug: PD patients H&Y=1.5-2 Medications OFF — Parkinson's patients will not take medications overnight prior to the study (20). Patients will perform both the stop-signal task and the go-only task. Experimental conditions will be counterbalanced across patients. This intervention will be given on a different day with respect to the Medication ON intervention. The order of intervention will be counterbalanced across subjects
  Arms: PD patients H&Y=1.5-2 Medications OFF
Behavioral: Healthy age-matched controls — Healthy controls will perform the stop signal task and the go-only task in the same day. The order of administration will be counterbalanced.
  Arms: Healthy age-matched controls
Drug: PD patients H&Y=3 Medications OFF — Parkinson's patients will not take medications overnight prior to the study (20). Patients will perform both the stop-signal task and the go-only task. Experimental conditions will be counterbalanced across patients. This intervention will be given on a different day with respect to the Medication ON intervention. The order of intervention will be counterbalanced across subjects
  Arms: PD patients H&Y=3 Medications OFF
Drug: PD patients H&Y=3 Medications ON — Parkinson's patients will be allowed to the first-morning dose of levodopa medicament (levodopa, dopamine agonists, anticholinergic drugs, or a combination of levodopa and an anticholinergic drug) which normally allowed the patient to attain the best control of symptoms one hour before being tested (19). Patients will perform both the stop-signal task and the go-only task. Experimental conditions will be counterbalanced across patients.
  Arms: PD patients H&Y=3 Medications ON

SUMMARY:
The effect of Levodopa medication on inhibitory control in Parkinson's patients is extremely debated despite the fact that this has potential clinical and therapeutic implications. A key confounding factor of many previous studies is that they did not take the disease duration in consideration. In fact, in moderate-to-advanced stages of Parkinson dopaminergic drugs could not produce a clear effect because too few dopaminergic cells for the drugs to operate on survived. Hence, in this study, we will compare the performance in the stop signal task in early-stage versus moderate-to-advanced stages Parkinson's patients both in ON and in OFF medication. In addition, to have a baseline measure of inhibitory control we will compare patient's performances with that of age-matched subjects.

DETAILED DESCRIPTION:
The ability to stop a pending action is fundamental for survival in a natural environment where events cannot be fully predicted. Sudden events, such as the appearance of a physical obstacle, often require a quick change of the planned motor strategy and the first step toward this goal is to suppress the pre-programmed actions. Thus voluntary inhibition plays a crucial role in cognitive control and behavioral flexibility (1, 2). It has been shown that Parkinson's patients suffer from a specific deficit in this functions (3, 4, 5). However, it is extremely debated whether and how Levodopa medication (levodopa, dopamine agonists, anticholinergic drugs, or a combination of levodopa and an anticholinergic drug) affects response inhibition. A number of studies measuring inhibitory control via the stop signal task in Parkinson's patients seem to indicate that dopaminergic medications do not influence this executive function (5, 6, 7). However, a recent study (8) found that Levodopa medication does not affect specifically inhibitory control or movement readiness, but the balance between them. In fact, Parkinson's patients in the OFF medication state were able to maintain response latencies in the same range as healthy controls, but they showed a significant reduction in the ability to stop reactions abruptly. In contrast, patients' performance shifted significantly when taking dopaminergic medications. They move slower but stopping improved relative to the off dopamine state. This pattern suggests a role for dopamine in modulating the tradeoff between the two action control processes. In addition, studies of other specific populations and healthy adults suggest that dopaminergic medications deserve reconsideration in response inhibition. For instance, positron emission (PET) studies have found that higher levels of striatal D1 and D2/D3 receptor availability predict better performance on the stop signal task (9, 10) and that response inhibition performance evokes dopamine release in prefrontal, parietal, and temporal cortex in healthy adults (11). Even more importantly, a few recent studies provided evidence that early-stage Parkinson's patients with response inhibition impairment seem to beneﬁt from dopaminergic treatment (12,13). Therefore, a plausible hypothesis is that the absence of a clear effect of dopaminergic medications could be ascribed to the fact that in most previous studies included Parkinson's patients in the moderate-to-advanced stages. In those patients, the diminished efﬁcacy of dopaminergic drugs could be a consequence that too few dopaminergic cells for the drugs to operate on survived (14).

Hence, the aim of the present work is to re-assess the impact of dopaminergic medications on inhibitory control on Parkinson's patients using a reaching version of the stop signal task (e.g. 4, 15, 16, 17, 18) taking the disease duration in consideration. To this aim, the investigators will compare the performance in the stop signal task in early-stage versus moderate-to-advanced stages Parkinson's patients both in ON and in OFF medication. Finally, to have a baseline measure of inhibitory control the investigators will compare patients' performances with those of age-matched subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handedness (as assessed by the Edinburgh Handedness Inventory)
2. Being in stable treatment with the administration of L-dopa and dopamine agonists (i.e. not having motor fluctuations and/or dyskinesia)
3. Having a Hoehn & Yahr score between 1.5 and 3

Exclusion Criteria:

1. Presence of severe sensory deficits
2. Presence of overt signs of dementia (a. mini-mental state examination, MMSE must be ≥24; b. intelligence quotient ≥75).
3. Comorbidity with other psychiatric disorders that might interfere with task execution (i.e. attentional disorders).
4. Presence of severe tremor or rigidity of the right arm in the OFF medication state.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Changes of length of the Stop Signal Reaction Time | Up to one year
  Reactive inhibition refers to the ability of a subject to react to the stop instruction, and it is measured by the stop-signal reaction time (SSRT). This variable cannot be measured, but it can be estimated by using the race model (21, 4, 16, 17, 18, 22).
Changes of the length of Reaction Times and Movement Times | Up to one year
  Proactive inhibition refers to the ability of subjects to shape their response strategy in anticipation of known task demands driven by endogenous signals. In the case of the countermanding task, the endogenous signal is represented by the awareness of the fact that sometimes an imperative stop-signal could have been presented. Proactive control could be assessed by measuring reaction times (i.e. the time to initiate a response, RTs) and movement times (i.e. the time to execute the motor response, MTs) of no-stop trials. Previous research has shown that when a movement is produced in the context of the countermanding task, that is when the subject executes a no-stop trial, its RT is lengthened (e.g. 4, 15, 16, 17, 18, 22) and its MT is shortened compared to situations in which the same movement has to be performed in the context of a simple RT-task (go-only trial; 4, 15, 17)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Neuromed Hospital, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirabella G. Should I stay or should I go? Conceptual underpinnings of goal-directed actions. Front Syst Neurosci. 2014 Nov 3;8:206. doi: 10.3389/fnsys.2014.00206. eCollection 2014. PMID 25404898
- [Background] Mirabella G, Lebedev Mcapital A, Cyrillic. Interfacing to the brain's motor decisions. J Neurophysiol. 2017 Mar 1;117(3):1305-1319. doi: 10.1152/jn.00051.2016. Epub 2016 Dec 21. PMID 28003406
- [Result] Gauggel S, Rieger M, Feghoff TA. Inhibition of ongoing responses in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Apr;75(4):539-44. doi: 10.1136/jnnp.2003.016469. PMID 15026491
- [Result] Mirabella G, Fragola M, Giannini G, Modugno N, Lakens D. Inhibitory control is not lateralized in Parkinson's patients. Neuropsychologia. 2017 Jul 28;102:177-189. doi: 10.1016/j.neuropsychologia.2017.06.025. Epub 2017 Jun 22. PMID 28647437
- [Result] Obeso I, Wilkinson L, Jahanshahi M. Levodopa medication does not influence motor inhibition or conflict resolution in a conditional stop-signal task in Parkinson's disease. Exp Brain Res. 2011 Sep;213(4):435-45. doi: 10.1007/s00221-011-2793-x. Epub 2011 Jul 28. PMID 21796541
- [Result] Claassen DO, van den Wildenberg WP, Harrison MB, van Wouwe NC, Kanoff K, Neimat JS, Wylie SA. Proficient motor impulse control in Parkinson disease patients with impulsive and compulsive behaviors. Pharmacol Biochem Behav. 2015 Feb;129:19-25. doi: 10.1016/j.pbb.2014.11.017. Epub 2014 Nov 29. PMID 25459105
- [Result] George JS, Strunk J, Mak-McCully R, Houser M, Poizner H, Aron AR. Dopaminergic therapy in Parkinson's disease decreases cortical beta band coherence in the resting state and increases cortical beta band power during executive control. Neuroimage Clin. 2013 Aug 8;3:261-70. doi: 10.1016/j.nicl.2013.07.013. eCollection 2013. PMID 24273711
- [Result] Wylie SA, van Wouwe NC, Godfrey SG, Bissett PG, Logan GD, Kanoff KE, Claassen DO, Neimat JS, van den Wildenberg WPM. Dopaminergic medication shifts the balance between going and stopping in Parkinson's disease. Neuropsychologia. 2018 Jan 31;109:262-269. doi: 10.1016/j.neuropsychologia.2017.12.032. Epub 2017 Dec 19. PMID 29269306
- [Result] Ghahremani DG, Lee B, Robertson CL, Tabibnia G, Morgan AT, De Shetler N, Brown AK, Monterosso JR, Aron AR, Mandelkern MA, Poldrack RA, London ED. Striatal dopamine D(2)/D(3) receptors mediate response inhibition and related activity in frontostriatal neural circuitry in humans. J Neurosci. 2012 May 23;32(21):7316-24. doi: 10.1523/JNEUROSCI.4284-11.2012. PMID 22623677
- [Result] Robertson CL, Ishibashi K, Mandelkern MA, Brown AK, Ghahremani DG, Sabb F, Bilder R, Cannon T, Borg J, London ED. Striatal D1- and D2-type dopamine receptors are linked to motor response inhibition in human subjects. J Neurosci. 2015 Apr 15;35(15):5990-7. doi: 10.1523/JNEUROSCI.4850-14.2015. PMID 25878272
- [Result] Albrecht DS, Kareken DA, Christian BT, Dzemidzic M, Yoder KK. Cortical dopamine release during a behavioral response inhibition task. Synapse. 2014 Jun;68(6):266-74. doi: 10.1002/syn.21736. Epub 2014 Feb 28. PMID 24677429
- [Result] Costa A, Peppe A, Mazzu I, Longarzo M, Caltagirone C, Carlesimo GA. Dopamine treatment and cognitive functioning in individuals with Parkinson's disease: the "cognitive flexibility" hypothesis seems to work. Behav Neurol. 2014;2014:260896. doi: 10.1155/2014/260896. Epub 2014 Jan 30. PMID 24825952
- [Result] van Wouwe NC, Kanoff KE, Claassen DO, Spears CA, Neimat J, van den Wildenberg WP, Wylie SA. Dissociable Effects of Dopamine on the Initial Capture and the Reactive Inhibition of Impulsive Actions in Parkinson's Disease. J Cogn Neurosci. 2016 May;28(5):710-23. doi: 10.1162/jocn_a_00930. Epub 2016 Feb 2. PMID 26836515
- [Result] Manza P, Amandola M, Tatineni V, Li CR, Leung HC. Response inhibition in Parkinson's disease: a meta-analysis of dopaminergic medication and disease duration effects. NPJ Parkinsons Dis. 2017 Jul 7;3:23. doi: 10.1038/s41531-017-0024-2. eCollection 2017. PMID 28702504
- [Result] Mirabella G, Iaconelli S, Modugno N, Giannini G, Lena F, Cantore G. Stimulation of subthalamic nuclei restores a near normal planning strategy in Parkinson's patients. PLoS One. 2013 May 3;8(5):e62793. doi: 10.1371/journal.pone.0062793. Print 2013. PMID 23658775
- [Result] Mirabella G, Iaconelli S, Romanelli P, Modugno N, Lena F, Manfredi M, Cantore G. Deep brain stimulation of subthalamic nuclei affects arm response inhibition in Parkinson's patients. Cereb Cortex. 2012 May;22(5):1124-32. doi: 10.1093/cercor/bhr187. Epub 2011 Aug 1. PMID 21810782
- [Result] Mirabella G, Pani P, Ferraina S. Context influences on the preparation and execution of reaching movements. Cogn Neuropsychol. 2008 Oct-Dec;25(7-8):996-1010. doi: 10.1080/02643290802003216. PMID 19378414
- [Result] Mirabella G, Pani P, Ferraina S. Neural correlates of cognitive control of reaching movements in the dorsal premotor cortex of rhesus monkeys. J Neurophysiol. 2011 Sep;106(3):1454-66. doi: 10.1152/jn.00995.2010. Epub 2011 Jun 22. PMID 21697448
- [Result] Mirabella G, De Vita P, Fragola M, Rampelli S, Lena F, Dilettuso F, Iacopini M, d'Avella R, Borgese MC, Mazzotta S, Lanni D, Grano M, Lubrani S, Modugno N. Theatre Is a Valid Add-On Therapeutic Intervention for Emotional Rehabilitation of Parkinson's Disease Patients. Parkinsons Dis. 2017;2017:7436725. doi: 10.1155/2017/7436725. Epub 2017 Nov 22. PMID 29359066
- [Result] Moro E, Scerrati M, Romito LM, Roselli R, Tonali P, Albanese A. Chronic subthalamic nucleus stimulation reduces medication requirements in Parkinson's disease. Neurology. 1999 Jul 13;53(1):85-90. doi: 10.1212/wnl.53.1.85. PMID 10408541
- [Result] Mirabella G, Pani P, Pare M, Ferraina S. Inhibitory control of reaching movements in humans. Exp Brain Res. 2006 Sep;174(2):240-55. doi: 10.1007/s00221-006-0456-0. Epub 2006 Apr 25. PMID 16636792
- [Result] Logan GD, Cowan WB, Davis KA. On the ability to inhibit simple and choice reaction time responses: a model and a method. J Exp Psychol Hum Percept Perform. 1984 Apr;10(2):276-91. doi: 10.1037//0096-1523.10.2.276. PMID 6232345